CLINICAL TRIAL: NCT00883012
Title: Immunogenicity, Safety and Efficacy of Influenza Vaccine in HIV Infected Children
Brief Title: Influenza Vaccine in HIV Infected Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Michelle Groome, Investigator, University of Witwatersrand, South Africa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Paediatric influenza vax
Record Dates: First submitted 2009-04-15; First posted 2009-04-17 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Influenza With Pneumonia, Influenza Virus Identified
Keywords: Viral-confirmed
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Influenza vaccine (Experimental): Two doses of trivalent sub-unit influenza vaccine (2009) to be administered one month apart
  Interventions: Biological: Trivalent sub-unit influenza vaccine
- Placebo (Placebo Comparator): Two doses of saline administered one month apart
  Interventions: Biological: Saline, 0.5ml

INTERVENTIONS:
Biological: Trivalent sub-unit influenza vaccine — Composition per 0.5 ml dose:
  Active substance:
  Split Influenza virus*, inactivated Strains for 2009 Southern hemisphere A/Brisbane/59/2007- like (H1N1) 15 micrograms**, A/Brisbane/10/2007 (H3N2) - like strain (A/Brisbane/10/2007 (IVR-147) 15 micrograms**, B/Florida/4/2006 - like strain (B/Brisbane/3/2007)15 micrograms** Two doses, one month apart
  Arms: Influenza vaccine
Biological: Saline, 0.5ml — Saline IMI, 0.5ml. Two doses one month apart
  Arms: Placebo

SUMMARY:
Influenza associated pneumonia causes significant morbidity in young HIV-infected children. Although annual vaccination against influenza is recommended for HIV infected children, it has not been implemented as routine care, due to the lack of data on disease burden and vaccine efficacy.

This study aims at determining the effectiveness of influenza vaccination in HIV infected children in South Africa.

DETAILED DESCRIPTION:
Influenza virus infects 30 to 50% of children under five years of age during the course of any epidemic. The attack rates of influenza virus associated illness during infancy remains high, and at least 50% of influenza associated hospitalisation amongst children occurs in infants <6 months of age. Approximately 33% of children would have been infected at least once during their first year of life. The estimated attack rates in children aged 0-5 and 6-12 months for influenza illness is 12.4/100 and 20.3/100 child years respectively. Influenza virus causes LRTI amongst 89% of children infected in the 6-12 month age group. The risk of influenza infection is higher amongst older children (2-5 years of age); however, the risk of developing LRTI (78 versus 2.5 per 100 child years) is greater amongst younger children (< 2 years of age).

In South Africa, the burden of influenza associated pneumonia has been characterized in HIV infected children. The incidence of severe pneumonia in which influenza virus was identified was 8.03 fold (95%CI 5.05-12.76) greater in HIV infected compared to HIV non-infected children (1 268 versus 148 per 100 000 child years) aged < 2 years. These rates however provide a very conservative estimate as to the burden of influenza illness, since it excludes children with influenza illness that were hospitalized for syndromes other than pneumonia as well as children managed as outpatients. Furthermore, although the duration of hospitalization for influenza associated pneumonia was similar between HIV infected and HIV uninfected children (median 4-5 days), there was a statistically non-significant increased risk of mortality among HIV infected children (8.0% versus 2.2%; P=0.20). Much of the differences in morbidity and mortality in HIV infected individuals with influenza-associated pneumonia may be due to contribution of other co-existing pathogens.

Recommendations made by the Advisory Committee on Immunization Practices (ACIP) advocating the annual use of the subunit influenza vaccine in HIV-1 infected children are largely founded on the theoretical concern regarding the potential severity of influenza disease in HIV-1 infected children. Although vaccination with the subunit influenza vaccine is recommended for HIV-1 infected children >6 months of age, there are concerns regarding the benefits of vaccination in these children. These include that in addition to a poor immune response to the vaccine, particularly in severely immunocompromised HIV-1 infected children, increases in plasma HIV RNA following vaccination have been described. The increase in plasma HIV RNA was transient and does not appear to be of any long-term clinical significance. Recently a few studies, with partly conflicting results, have been undertaken evaluating the immunogenicity of influenza vaccination in children on antiretroviral therapy. However, no such studies have been undertaken in Africa or Asia where the burden of paediatric HIV is the greatest.

The routine use of influenza vaccine in HIV infected children remains low, partly related to the lack of adequate data regarding the burden of influenza associated disease in these children as well as the lack on any vaccine-efficacy data in HIV infected children. Determining the burden of disease and effectiveness of influenza vaccine in HIV infected children will have a bearing on routine immunization recommendations as well as planning for future influenza pandemics.

Differences in the epidemiology of HIV between developing and developed countries in which the prevalence of HIV is low to that of high-burden sub-Saharan African countries makes it necessary to be cautious in extrapolating data and recommendations of developed countries to developing countries. These differences may include: i. differences in standard of care, including access to prophylaxis against opportunistic infections and use of highly active anti-retroviral therapy (HAART); ii. differences in risk for disease from opportunistic pathogens, e.g. Mycobacterium tuberculosis, etc. These differences may all contribute to differences in the risk and severity of influenza illness among HIV infected individuals from these communities as well as possibly responsiveness and effectiveness of vaccination.

It is within this context that this study aims at determining the effectiveness of influenza vaccination in HIV infected children in South Africa. The significance of the findings from this study will help quantify the burden of influenza illness in African HIV infected children, in the era of HAART, as well as assist in making more informed recommendations for the use of influenza vaccine in HIV infected children and in guiding national policy for preparing for a future influenza virus-pandemic.

350 Patients will be recruited at Chris Hani-Baragwanath Hospital, Soweto, South Africa onto this prospective, double-blind, placebo randomised controlled trial evaluating the efficacy of a tri-valent sub-unit influenza vaccine in HIV infected children. Participants will be randomized to receive either two doses of Influenza sub-unit vaccine or placebo one month apart, preceding the 2009 Influenza season. 100 children will be included into the immunogenicity cohort, and have blood drawn to evaluate baseline influenza strain specific antibody levels and subsequent levels one-month following the first and second doses of study vaccine.

Study participants will be followed up during the course of the influenza season, which will be defined as starting 1st May 2009 and ending 30th September 2009. Subjects will be contacted weekly to determine whether they fulfill the criteria for Influenza-like illness. Subjects who fulfill the criteria for diagnosing ILI will be requested to come into the clinic within 48 hours for further investigation, which will involve a nasopharyngeal aspirate (for identification of respiratory viruses), nasopharyngeal swab (for identification of Streptococcus pneumoniae colonization) and blood draw (for culture and Streptococcus pneumoniae testing).

ELIGIBILITY:
Inclusion Criteria:

* HIV infected children with CD4% ≥ 15% performed within the previous 3 months in relation to the date of randomization.
* Age 6 month- 5 years old.
* Willing and able to maintain weekly contact at least during period of April - August (i.e. presupposed influenza period) either through SMS or telephonic contact.
* Willing and able to adhere to study protocol re: attendance to clinic for scheduled and illness visits.

Exclusion Criteria:

* Any contraindication to influenza vaccination, including known allergy to egg.
* History of chronic lung disease which required maintenance therapy either currently or in the past 6 months.
* Any contraindication to intramuscular injections.
* Current known grade 3 or grade 4 laboratory or clinical toxicity as per DAIDS toxicity tables.
* Any previous history of influenza vaccination.
* Plan to emigrate from the study area within the next year.
* On steroid therapy for > 21 days (current or within the past 30 days).
* In the investigators opinion unable to maintain study procedures.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 412 (Actual)
Dates: Start 2009-02; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of a tri-valent influenza sub-unit vaccine, in HIV infected children with a CD4+ percentage >15% against vaccine-strain viral confirmed influenza illness. | One year
Define the immunogenicity of influenza vaccination in a nested cohort of HIV infected children with CD4+ percentage >15% that are naïve to anti-retroviral or on antiretroviral therapy for more than 3 months | One year

SECONDARY OUTCOMES:
Determine the safety of influenza vaccination in relation to solicited vaccine-related adverse events in the 72 hour period post-vaccination and any other unsolicited adverse event. | One year
Compare the effect of the influenza vaccination on viral control and CD4+ cell count in HIV infected children six months following influenza vaccination. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Shabir A Madhi, MD, PhD, Principal Investigator — VPD- RMPRU
Locations (1):
- Chris Hani Baragwanath Hospital, Soweto, Gauteng, South Africa